CLINICAL TRIAL: NCT00927628
Title: Incidence and Factors Related to Macular Hole Reopening
Brief Title: Macular Hole Reopening
Status: Completed | Type: Observational
Sponsor: Shinjo Ophthalmologic Institute (Other)
Responsible Party: Dr. Kazuyuki Kumagai, Shinjo Ophthalmologic Institute
Other Study IDs: ShinjoOI
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Vitrectomy
Keywords: vitrectomy; macular hole; ILM peeling
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vitrectomy: Patients underwent vitrectomy with or without internal limiting membrane (ILM) peeling for an idiopathic full-thickness macular hole. Simultaneous phacoemulsification with intraocular lens implantation was performed on all phakic patients who were >40-years-of-age.
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Patients underwent vitrectomy with or without internal limiting membrane (ILM) peeling for an idiopathic full-thickness macular holes. Simultaneous phacoemulsification with intraocular lens implantation was performed on all phakic patients who were >40-years-of-age.

SUMMARY:
The purpose of this investigation was to determine the incidence and the factors that cause a reopening of a macular hole (MH) after a surgical closure.

DETAILED DESCRIPTION:
A reopening of a macular hole (MH) is a well-known complication of successfully closed MHs. Recently, internal limiting membrane (ILM) peeling has become widely used as an adjunctive procedure during MH surgery. The incidence of a reopening of a MH is 0 to 8.6% in eyes in which the ILM was peeled off, and 2 to 16% in which the ILM was not peeled off. Part of the variation in the percentages of reopening was the length of the follow-up period; eyes with longer follow-up periods have higher incidences of reopening.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent vitrectomy with or without internal limiting membrane (ILM) peeling for an idiopathic full-thickness macular hole

Exclusion Criteria:

* eyes with previous vitreous surgery, cystoid macular edema from any cause, and traumatically-induced MH were excluded.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eight hundred seventy-seven eyes of 831 patients with a mean age of 64.9 ± 8.0 years were studied.
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 1990-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
A complete clinical examination including BCVA, slit-lamp biomicroscopy with a contact lens, indirect ophthalmoscopy, and fundus photography were performed post surgery. | Patients were examined preoperatively and postoperatively on day one, and at two weeks, and one, three, and six months. Thereafter, they were examined every three to six months.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuyuki Kumagai, MD, Principal Investigator — Shinjo Ophthalmologic Institute
Locations (1):
- Shinjo Ophthalmologic Institute, Miyazaki, Miyazaki, Japan

REFERENCES:
- [Background] Duker JS, Wendel R, Patel AC, Puliafito CA. Late re-opening of macular holes after initially successful treatment with vitreous surgery. Ophthalmology. 1994 Aug;101(8):1373-8. doi: 10.1016/s0161-6420(13)31174-9. PMID 8058282
- [Background] Kokame GT. Recurrence of macular holes. Ophthalmology. 1995 Feb;102(2):172-3. doi: 10.1016/s0161-6420(95)31042-1. No abstract available. PMID 7862400
- [Background] Kumagai K, Furukawa M, Ogino N, Uemura A, Demizu S, Larson E. Vitreous surgery with and without internal limiting membrane peeling for macular hole repair. Retina. 2004 Oct;24(5):721-7. doi: 10.1097/00006982-200410000-00006. PMID 15492625
- [Background] Gross JG. Late reopening and spontaneous closure of previously repaired macular holes. Am J Ophthalmol. 2005 Sep;140(3):556-8. doi: 10.1016/j.ajo.2005.03.044. PMID 16139019
- [Background] Kumagai K, Furukawa M, Ogino N, Larson E, Uemura A. Long-term outcomes of macular hole surgery with triamcinolone acetonide-assisted internal limiting membrane peeling. Retina. 2007 Nov-Dec;27(9):1249-54. doi: 10.1097/IAE.0b013e3180ed45cc. PMID 18046233
- [Background] Kumagai K, Ogino N, Furukawa M, Larson E, Uemura A. Surgical outcomes for patients who develop macular holes after pars plana vitrectomy. Am J Ophthalmol. 2008 Jun;145(6):1077-80. doi: 10.1016/j.ajo.2008.01.030. Epub 2008 Apr 18. PMID 18378210